CLINICAL TRIAL: NCT06159166
Title: A Phase 1/2a Open-label, Multicenter Dose Finding Study to Evaluate the Safety and Anti-tumor Activity of Mirdametinib Monotherapy in Adults With Neurofibromatosis 1 (NF1) and Cutaneous Neurofibromas (cNF).
Brief Title: Mirdametinib Monotherapy in Adults With Neurofibromatosis 1 (NF1) and Cutaneous Neurofibromas (cNF).
Acronym: Mirda
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Neurofibromatosis Therapeutic Acceleration Program (Unknown); SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00365255; J23129 (Other: SKCCC)
Record Dates: First submitted 2023-11-08; First posted 2023-12-06 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: NF1; Cutaneous Neurofibroma; Monotherapy
Keywords: Mirdametinib
MeSH Terms: interventions — mirdametinib

STUDY DESIGN:
Intervention Model Description: Phase 1 will test the safety of multiple dose regimens of mirdametinib, in order to identify a recommended phase 2 dose(s) for phase 2a. The phase 1 portion will enroll participants in dose regimens 1 to 3 concurrently. Enrollment of participants to dose regimen 4 will be conducted only if no DLT occurred in any of the three previous regimens within at least, the first three cycles. The study will continue until one of the following stopping conditions is met.
  * The RP2D(s) have been identified with sufficient accuracy (The dose regimen(s) selected as the RP2D have been fully enrolled with at least 3 cycles of treatment completed for all participants)
  * All dose regimens are deemed to have unacceptable safety
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): For the Phase 1 portion, treatment will be administered continuously (Dose regimens 1, 2, 4) or intermittently (Dose regimen 3; 3 weeks on/1 week off) in 28-day cycles). All participants will receive study drug until:
  1. cessation of study treatment due to death, intolerance, or withdrawal of consent from the study;
  2. completion of 24 cycles of treatment (unless the investigator's benefit-risk assessment supports continued treatment);
  3. participants enroll in the phase 2a portion of the study;
  4. disease progression; or
  5. Investigator's decision.
  Treatment period ends with the administration of the last dose. The study ends 30 days after the last dose
  Interventions: Drug: Mirdametinib
- Phase 2 (Experimental): For the Phase 2 portion, treatment will be administered based on recommended RP2D from Phase 1. All participants will receive study drug until:
  1. cessation of study treatment due to death, intolerance, or withdrawal of consent from the study;
  2. completion of 24 cycles of treatment (unless the investigator's benefit-risk assessment supports continued treatment;
  3. disease progression; or
  4. Investigator's decision.
  Treatment period ends with the administration of the last dose. The study ends 30 days after the last dose.
  Interventions: Drug: Mirdametinib

INTERVENTIONS:
Drug: Mirdametinib — This study is designed to assess Mirdametinib safety and efficacy in two phases: phase 1 tests the safety of up to four dose regimens of Mirdametinib, administered continuously or intermittently (3 weeks on/1 week off) to identify up to two recommended phase 2 doses. Phase 2a of the study will test the safety and efficacy of the recommended phase 2 dose(s) in adults with NF1 and cNF. The following dosing strategy will be assessed in participants ≥ 18 years old with NF1 and a minimum of 12 measurable cNF who desire systemic treatment of their cNF due to disfigurement, pain or itching. Each treatment cycle in this study is 28 days.treatment cycle in this study is 28 days.

SUMMARY:
This is a Phase 1/2a, open-label, non-randomized, multi-dose study of mirdametinib monotherapy in adults with NF1 and cNF.

In both Phases of the study, participation in the study will comprise three periods: screening, treatment and post-study safety follow-up to be performed at the NF1 and cNF specialty center: Johns Hopkins University.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, non-randomized, multi-dose study of mirdametinib monotherapy in adults with NF1 and cNF. The study will be conducted in two phases:

Phase 1 will test the safety of multiple dose regimens of mirdametinib, in order to identify a recommended phase 2 dose(s) for phase 2a. The phase 1 portion will enroll participants in dose regimens 1 to 3 concurrently. Enrollment of participants to dose regimen 4 will be conducted only if no dose limiting toxicities (DLT) occurred in any of the three previous regimens within at least, the first three cycles. The study will continue until one of the following stopping conditions is met.

* The RP2D(s) have been identified with sufficient accuracy. The dose regimen(s) selected as the RP2D have been fully enrolled with at least 3 cycles of treatment completed for all participants)
* All dose regimens are deemed to have unacceptable safety

Phase 2a of the study will test the efficacy and safety of a maximum of two RP2Ds in adults with NF1 and cNF.

This study will be considered complete once all participants have ceased study treatment due to death, disease progression, intolerance, withdrawal of consent from the study, physician discretion, or completed a maximum of 48 cycles of treatment across both phase 1 and phase 2a. Each treatment cycle is 28 days.

In both Phases of the study, participation in the study will comprise three periods: screening, treatment and post-study safety follow-up to be performed at Johns Hopkins University.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for NF12
2. ≥ 18 years of age
3. Have a minimum of 24 measurable cNF (2 target areas of ≥6 measurable cNF)

   a. Measurable is defined as: i. non-pedunculated (no stalk) ii. surrounded by uninvolved skin and not adjacent to another cNF lesion iii. measuring ≥ 0.5 cm in the longest diameter and ≥ 0.5 cm in height iv. the 24 cNF must be located in two Target Areas. One target area must be located on the back and must have at least 6 measurable cNF. The second target area can be in any of the following body regions with at least 6 cNF: head and neck; upper extremities; anterior chest wall, anterior abdominal wall; pelvic region/gluteal region; lower extremities.
4. Participants must have cNF that meet eligibility criteria located within the two study designated target areas or outside of the target areas amenable to biopsy. If biopsy is taken within the target area there must be a minimum of 6 cNF remaining for long term surveillance after biopsy. Participants must be willing to undergo pre-, and on-treatment tumor biopsies providing fresh tumor tissue; there should be no contraindication for serial biopsy
5. Karnofsky performance level of ≥ 80%.
6. Adequate organ and bone marrow function as defined by the following Screening laboratory values:

   1. Absolute neutrophil count ≥ 1500 cells/µL;
   2. Platelets ≥ 100 x 103/µL;
   3. Hemoglobin ≥ 9.5 g/dL;
   4. Serum albumin ≥ 2.8 g/dL;
   5. Calculated creatinine clearance at Screening ≥ 60 mL/min (by Cockcroft-Gault formula) OR a normal serum creatinine.
7. Participant is willing and able to comply with all aspects of the protocol
8. Ability to understand and the willingness to sign written informed consent document(s).
9. Women of childbearing potential (WOCBP) must not be pregnant or breastfeeding during any portion of the study and must use an adequate method to avoid pregnancy during the study period and for 6 months after treatment conclusion and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during the study and for a period of 6 months after last dose of study treatment. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment (see the Approved Methods of birth control listed below).

   * In order for a woman to be determined not of childbearing potential, she must have ≥ 12 months of non-therapy-induced amenorrhea or be surgically or medically sterile.
   * WOCBP must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test result at the Baseline visit prior to the first dose of study treatment.

     * The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
10. Male participants are eligible to participate if they agree to the following during the treatment period and for at least 90 days after the last dose of study treatment:

    * Refrain from donating sperm

PLUS either:

* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent until 90 days after the last study drug treatment; OR
* Must agree to use a male condom when having sexual intercourse with a WOCBP and their female partner must utilize one the approved methods of birth control below:

Approved Methods of birth control for this study are:

* Total abstinence
* Male or female sterilization (vasectomy in males or surgical removal of ovaries or uterus in females)
* Unsterilized male study participants must use a male condom and their female partner must use one of the methods below:
* Unsterilized female study participants must use one of the following highly effective methods listed below:

Acceptable birth control methods which are considered highly effective if they result in a failure rate of less than 1% per year when used consistently and correctly:

* Combined (estrogen and progestogen containing) hormonal contraceptive that stops the release of eggs from the ovary (oral, intravaginal, or transdermal)
* Progestogen-only hormonal contraception that stops the release of eggs from the ovary (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion or bilateral tubal ligation

Exclusion Criteria:

1. Participant has a altered screening values:

   1. alanine transaminase (ALT) value of > 2.0 x upper limit of normal (ULN);
   2. total bilirubin value of > 1.5 x ULN (isolated bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%);
2. Participant has a history of malignancy associated hypercalcemia;
3. Participant has an active parathyroid disorder, hyperphosphatemia at Screening (serum phosphorus > 1 x ULN), or serum calcium (mg/dL) x serum phosphorus (mg/dL) product > 70 at Screening;
4. Any clinically significant active or known history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
5. Hepatitis serology will be tested at Screening. Participants who are hepatitis B surface antigen (HBsAg) positive or hepatitis C virus (HCV) antibody positive at Screening must not be enrolled until further definite testing with hepatitis B virus (HBV) deoxyribonucleic acid (DNA) titers is < 500 IU/mL or HCV ribonucleic acid (RNA) polymerase chain reaction test is negative;
6. Lymphoma, leukemia, or any malignancy (including malignant glioma or MPNST) within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years;
7. Breast cancer within the past 3 years;
8. Active optic glioma or other low-grade glioma requiring treatment with chemotherapy or radiation therapy.

   a. Participants not requiring treatment are eligible. Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study;
9. Abnormal QT interval corrected by Fridericia's formula (> 450 msec for male participants, > 470 msec for female participants, or > 480 msec for participants with known bundle branch block), calculated from triplicate ECG readings taken approximately 2 to 3 minutes apart and averaged at Screening;
10. Participant has experienced any of the following within 6 months (24 weeks) of signing informed consent/assent: clinically significant cardiac disease, myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism;
11. A recorded LVEF < 55% at screening or within 3 years of signing informed consent/assent, OR has a history of congestive heart failure;
12. Participants with a history of, or evidence of, retinal pathology on ophthalmologic examination that is considered a risk factor for central serous retinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration. Participants will be excluded from study participation if they have any of the following risk factors for RVO at Screening:

    * Intraocular pressure > 21 mmHg;
    * Serum cholesterol > 300 mg/dL;
    * Serum triglycerides > 300 mg/dL;
    * Hyperglycemia (fasting blood glucose > 125 mg/dL or random blood glucose > 200 mg/dL);
    * Hypertension (BP ≥ 140/90 mm Hg)
13. History of glaucoma;
14. Known history of a positive human immunodeficiency virus (HIV) antibody test;
15. Known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of mirdametinib (e.g., gastric bypass, lap band, or other gastric procedures). Delivery of mirdametinib via nasogastric tube or gastrostomy tube is not allowed.
16. Previously treated with MEK inhibitor including mirdametinib (PD-0325901) and had to stop treatment due to adverse event.
17. Currently receiving therapy with a MEK inhibitor including mirdametinib (PD-0325901) or treated with a MEK inhibitor in the 12 months prior to prior to first dose of study treatment.
18. Received radiation therapy within the 6 months prior to prior to first dose of study treatment. Participants who have received radiation to the orbit at any time are excluded.
19. Pregnant or breastfeeding women may not take study drug.
20. Current enrollment or past participation in any other clinical study (excluding observational studies) within 28 days of first dose of study treatment.
21. Known sensitivity to the study treatment, or components thereof, or drug or other allergy that, could compromise safety of the subject
22. Participant is receiving systemic (oral, inhaled, of IV/SC) or ocular glucocorticoid therapy (with the exception of participants with endocrine deficiencies who are allowed to receive physiologic or stress doses of steroids, if necessary) within 14 days prior to first dose of study treatment;
23. Participants are excluded if they have severe and/or uncontrolled medical disease or social situation, which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration, congestive heart failure, drug or alcohol dependence, etc.).
24. Participants is receiving systemic treatment of a pan-cytochrom 450 (CYP) inducers such as rifampin or ritonavir within 14-days prior to first dose of study treatment Drug Development and Drug Interactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of continuous and three week on-one week off dosing of mirdametinib in adults with NF1 and cutaneous neurofibromas (cNFs). | Up to 28 days
  Phase 1 will test the safety and tolerability of multiple dose regimens of mirdametinib, in order to identify the recommended phase 2 dose(s) for phase 2a. The study will continue until one of the stopping conditions is met.
  * The RP2D(s) have been identified with sufficient accuracy (The dose regimen(s) selected as the RP2D have been fully enrolled with at least 3 cycles of treatment completed for all participants)
  * All dose regimens are deemed to have unacceptable safety The study will continue until one of the following stopping conditions is met.
  * The RP2D(s) have been identified with sufficient accuracy (The dose regimen(s) selected as the RP2D have been fully enrolled with at least 3 cycles of treatment completed for all participants)
  * All dose regimens are deemed to have unacceptable safety
Define the recommended phase 2 dose (RP2D) of mirdametinib in adults with NF1 and cNF. | Up to 28 days
  Phase 2a of the study will test the efficacy and safety of a maximum of two RP2Ds in adults with NF1 and cNF.
• Evaluate the preliminary anti-tumor activity of mirdametinib monotherapy in adults with NF1 and cNFs. | Up to 28 days
  Evaluate the efficacy of mirdametinib monotherapy at the RP2D in adults with NF1 and cNF. We will determine efficacy of Anti-tumor activity with 3D photography (Sum of the surface area, sum of the tumor volume, sum of the longest diameter) and Digital Caliper (Sum of the longest diameter).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Romo, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States